CLINICAL TRIAL: NCT05026281
Title: Intérêt de l'Utilisation du "Quantra® Haemostasis Analyser" Lors de la Prise en Charge Des Patients présentant Une hémorragie Grave Sous Anticoagulant Oral
Brief Title: Bleeding Oral Anticoagulant Analyzer (BOA)
Acronym: BOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Hôpital Edouard Herriot (Other); University Hospital of Saint-Etienne (Other); University Hospital, Grenoble (Other); University Hospital, Tours (Other); Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AOI 2020 TEISSANDIER; 2020-A03240-39 (Other: ANSM)
Record Dates: First submitted 2021-08-13; First posted 2021-08-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2022-09

CONDITIONS: Anticoagulants and Bleeding Disorders
Keywords: Haemorrhage; Anticoagulant; Emergency; Quantra analyzer
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage; Emergencies

STUDY DESIGN:
Intervention Model Description: H0 : blood analyse with Quantra® H0+30 min : blood analyse with Quantra® D0+30 : end of study
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): at H0 and H0+30min = blood sample taken
  Interventions: Device: Quantra analyzer

INTERVENTIONS:
Device: Quantra analyzer — one additional tube will be collected during the usual blood test at two different time and analyzed by Quantra ®

SUMMARY:
The quality of the reversion of these serious hemorrhagic accidents under oral anticoagulants depends on the adequate use of reversion products but also on the speed of obtaining hemostasis data allowing to evaluate the effectiveness of this "chemical" hemostasis. .

Clot formation can be studied using different visco-elastic methodologies (thromboelastography or thromboelastometry) with a detectable change in clot formation with oral anticoagulants.

These techniques have been proven in patients who are often unstable and present with severe trauma with hemorrhagic shock, thus making it possible to guide the transfusion protocol. However, the level of recommendations in these patients, who are often polyhydrated and poly-transfused, is grade 1c due to small-scale studies with difficulty in analyzing the values of the visco-elasticity parameters in these patients. In addition, these methods are little used in current practice because of their difficult reading.

The use of visco-elastic methods in patients on oral anticoagulants has been little studied. However, taking an oral anticoagulant mainly causes coagulation disorders. The use of these methods would make it possible to assess the impact of the anticoagulant on hemostasis and to verify the correct reversion of hemostasis parameters. Quantra®, one of the visco-elastic methods, would make it possible to speed up the evaluation in the context of biology relocated to the patient's bed with a simplified reading of the factors involved in the formation of the clot in order to allow an immediate evaluation the quality of the reversion performed which may have an impact on the re-administration of reversion products or even an adaptation of the dose of reversion products according to the initial parameters at the time of severe bleeding before reversion. The objective of this pilot study is to study the metrological evolution, before and after reversion, of the hemostasis parameters evaluated by the Quantra® system from HemoSonics in a patient being his own control in the context of a severe hemorrhage occurring on oral anticoagulants (VKA or DOA).

DETAILED DESCRIPTION:
This multicenter, prospective, cohort pilot study of physiopathology and physio-pharmacology, testing the added value of innovative functional exploration in addition to routine monitoring, in patients eligible for urgent reversion from anticoagulant therapy.

This study is part of the patient's routine care without modifying his management. In fact, eligible patients with severe bleeding under oral anticoagulant therapy will be treated according to departmental habits. The study will only consist of the addition of the analysis of a blood sample using the Quantra® before and after reversion without modification of the management.

All patients will be followed for the duration of hospitalization.

Primary objective :

The objective of this pilot study is to study the behavior of viscoelastic hemostasis parameters assessed by the Quantra® System in the context of severe bleeding occurring under oral anticoagulants (VKA or DOA).

Secondary objectives :

To study the effect of reversion of oral anticoagulants on hemostasis parameters assessed by the Quantra® system in the context of severe bleeding.

To study, in the context of severe bleeding, the relationship between the hemostasis parameters assessed by the Quantra® system and:

* conventional hemostasis parameters,
* the severity of the bleeding events before reversion, in the context of severe bleeding,
* recurrent bleeding or thrombotic events occurring during hospitalization.

The primary endpoint will be all of the Quantra® parameter values measured during the patient's therapeutic monitoring (before and after) without prioritization. The parameters of Quantra® are:

* CT: Clotting time (in seconds)
* CTH: Clotting time with Heparinase (in seconds)
* CTR: CT / CTH ratio clotting time
* CS: overall stiffness of the clot (hPa)
* PCS: Contribution of platelets to clot stiffness (hPa) FCS: Contribution of fibrinogen to clot stiffness (hPa)

Secondary endpoints:

* Classic coagulation tests: (TP / INR), TCA, Fibrinogen, FII, FV, FVII, FX
* Drug concentration (for DOA) by dilute thrombin time or specific anti-Xa activity
* Type and volume of filling solutes before reversion
* Assessment of blood loss (Hb, size of the hematoma)
* Clinical outcome of reversion: haemostatic efficacy rate at 24 hours, occurrence of haemorrhagic or thrombotic recurrences during hospitalization
* Duration of hospitalization

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient, male or female, treated long term with an oral anticoagulant (anti-vitamin K or direct), admitted to a hospital emergency department for intracerebral, digestive or intramuscular hemorrhage, defined as major according to the criteria of the International Society of Thrombosis and Haemostasis1. These three sites of bleeding are the most common.
2. Capable of giving informed consent to participate in research or in the event of emergency care for a reference person.
3. Affiliated with a Social Security scheme.

Exclusion Criteria:

1. Incapable major.
2. Administration within the last 24 hours of parenteral anticoagulant.
3. Refusal of participation.
4. Pregnant or breast feeding mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
change in viscoelastic hemostasis parameters assessed by the Quantra® system in the context of severe bleeding occurring under oral anticoagulants (VKA or DOA) | Hour 0 and Hour 0+30min
  Quantra® parameters were measured during the patient's therapeutic monitoring (before and after) without prioritization. The parameters of Quantra® are:
  CT / CTH ratio clotting time overall stiffness of the clot (hPa) Contribution of platelets to clot stiffness (hPa) Contribution of fibrinogen to clot stiffness (hPa)
Change in viscoelastic hemostasis parameters assessed by the Quantra® system in the context of severe bleeding occurring under oral anticoagulants (VKA or DOA) | Hour 0 and Hour 0+30min
  Quantra® parameters were measured during the patient's therapeutic monitoring (before and after) without prioritization. The parameters of Quantra® are:
  CT : clotting time (in seconds) CTH clotting time with heparinase (in seconds)

SECONDARY OUTCOMES:
Coagulation test | Hour 0; Hour 0+30min; Hour 0+6 hours
  change in activated partial thromboplastin time (APTT) measures
Coagulation test | Hour 0; Hour 0+30min; Hour 0+6 hours
  change in prothrombin time test values
Coagulation test | Hour 0; Hour 0+30min; Hour 0+6 hours
  changes in levels of fibrinogen
Coagulation test | Hour 0; Hour 0+30min; Hour 0+6 hours
  change in Factor II assay
Coagulation test | Hour 0; Hour 0+30min; Hour 0+6 hours
  change in Factor V assay
Coagulation test | Hour 0; Hour 0+30min; Hour 0+6 hours
  change in Factor VII assay
Coagulation test | Hour 0; Hour 0+30min; Hour 0+6 hours
  change in Factor X assay
anti-factor Xa activity measurement | Hour 0; Hour 0+30min; Hour 0+6 hours
  change in anti-factor Xa activity measurement
Type of filling solutes before reversion | Hour 0
  Type of filling solutes before reversion
Volume of filling solutes before reversion | Hour 0
  Volume of filling solutes before reversion
Evaluation of blood loss | Hour 0
  haemoglobin concentration
Evaluation of blood loss | Hour 0
  haematoma size
Clinical haemostasis evolution | Hour 0+24
  haematoma volume
Clinical haemostasis evolution | Hour 0+24
  Haematoma pain on numeric scale (0-10 points)
Clinical issue of reversion | Hour 0+24
  efficacy haemostatic rate at 24 hours
Clinical issue of reversion | Hour 0+24
  Recurrence of bleeding during hospitalization
Duration of hospitalization | at the end of hospitalization
  how many days the patient is hospitalized
phone call | Month 0+1
  report of any adverse event occured in the month after the end of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Teissandier, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (6):
- France (6):
  - University Hospital, Clermont-Ferrand
  - Grenoble University Hospital, Grenoble
  - Edouard Herriot University Hospital, Lyon
  - La Pitié-Salpétrière, Paris
  - Saint Etienne University Hospital, Saint-Etienne
  - Tours University Hospital, Tours